CLINICAL TRIAL: NCT03581604
Title: Diagnostic De-labeling of Patients With False Diagnosis of Penicillin Allergy: A Tool for Improving Antimicrobial Treatment and Reducing Antimicrobial Resistance
Brief Title: De-labeling of Patients With False Diagnosis of Penicillin Allergy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Eva Stylianou, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/2119/REK
Record Dates: First submitted 2018-05-04; First posted 2018-07-10 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Allergy Drug
Keywords: Penicillin/b-lactams
MeSH Terms: conditions — Drug Hypersensitivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Patient group consisting of patients labeled as penicillin allergic.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients labeled as penicillin allergic (Other): Patients labeled as penicillin allergic will be allergologically investigated to confirm/exclude the diagnosis. Allergy work-up will be performed. Blood samples will be obtained.Questionnaire to evaluate the effectiveness of the intervention.
  Interventions: Diagnostic Test: Allergy work-up; Other: Blood samples

INTERVENTIONS:
Diagnostic Test: Allergy work-up — Allergy work-up
Other: Blood samples — Blood samples

SUMMARY:
The purpose of this study is to estimate the prevalence of penicillin allergy, evaluate the diagnostic value of the allergologic work-up used in the study, and the health effects of penicillin allergy.

DETAILED DESCRIPTION:
Penicillin allergy is the most common of self-reported drug allergies and un-verified penicillin allergy is a significant and growing public health problem. 10% of all patients report penicillin allergy. However, there is large discrepancy between reported penicillin allergy and true allergy. Despite its high prevalence, greater than 90% of such patients are in fact able to tolerate the medication without allergic reactions.

In this study patients having a penicillin allergy label will be investigated to confirm or to exclude the allergy diagnosis. The diagnostic value of the allergen test panel and the allergologic work-up will be evaluated. Clinical parameters as well as immunological will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are referred to the department of Pulmonary medicine with clinical history suspected of having penicillin allergy.
* The control group will be healthy adult volunteers with no history of any personal or family history of drug allergy, atopy, inflammatory or autoimmune diseases.

Exclusion Criteria:

* Systemic reactions such as DRESS, any internal organ involvement
* Clinical history of Type II-III hypersensitivity reaction
* Severe Type IV hypersensitivity reaction such as Stevens-Johnson syndrome, toxic epidermal necrolysis, DRESS, vasculitis, acute generalized exanthematous pustulosis
* Chronic idiopathic urticaria on antihistamine maintenance treatment/anti-IgE treatment
* Medication which can affect the test outcome
* Active signs of an underlying disease such as uncontrolled asthma
* Cardiac disease with increased risk of serious anaphylaxis
* Pregnancy/Breastfeeding
* Reaction within the last 4-6 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Penicillin allergy in the studied group | up to 4 years
  Frequency of true penicillin allergy in the study group
Negative predictive value of the allergy work- up | 3 weeks
  If the allergy work-up is negative, drug provocation test with penicillin will be performed. The purpose of the drug challenge is to confirm lack of allergy and confirm the negative predictive value of the allergy work-up.

SECONDARY OUTCOMES:
Use of b-lactams after negative allergy work-up and development of new drug reactions following negative testing. | 12 months
  Patients going through an allergy workup with negative results, will be retrospectively contacted within one year after investigation. Telephone interview where the following questions will be asked:1) "Have you received antibiotic therapy since being seen in the allergy clinic?" 2) "If you have been treated, what drug did you take?" 3) "As a result of this, did you have a reaction to the antibiotics?" "If yes, what kind of reaction have you developed?" 4) "If you didn't take the drug you were challenged with what was the reason for that?"

CONTACTS AND LOCATIONS:
Overall Officials: Eva Stylianou, Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Dpt of Pulmonary Diseases, Ullevål, Oslo, Postbox 4950 Nydalen, Norway